CLINICAL TRIAL: NCT00579228
Title: Vascular Risk Progression in Normal and Diabetes Control Subjects
Brief Title: Vascular Risk Progression in Normal and Diabetic Control Subjects.
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0124-07-EP
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Diabetes; Inflammation
Keywords: Diabetes; Vascular risk; Inflammation
MeSH Terms: conditions — Diabetes Mellitus; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1 Cardiovascular disease (CVD) in Participants without diabetes: Progression of cardiovascular disease (CVD) in participants without diabetes
- 2 Cardiovascular disease (CVD) in participants with type 2 Diabetes: Progression of cardiovascular disease (CVD) in participants with type 2 Diabetes with good control
- 3 Cardiovascular disease (CVD) in participants with type 1 diabetes: Progression of cardiovascular disease (CVD) in participants with type 1 diabetes with good control

SUMMARY:
The purpose of this study is to look at the progression of cardiovascular disease (CVD) in normal control individuals and in patients with controlled diabetes.

DETAILED DESCRIPTION:
Cardiovascular disease remains the greatest cause of mortality in people with diabetes mellitus. This observation study will evaluate non-traditional risk factors for their contributions to vascular disease progression as determined by carotid intima media thickness and history of vascular disease events over 1 year. This study requires annual checks of blood, urine, history, and carotid ultrasound for carotid intimal medical thickness.

ELIGIBILITY:
Inclusion Criteria:

* 19 years old or more and willing to return for annual testing for 2 years.
* Those with Diabetes need to have the condition for at least 5 years.
* Normal controls need to have no diabetes, kidney disease, or chronic disease.

Exclusion Criteria:

* Estimated GFR <60 (mL/min/1.73m2)
* Any condition that would change weight dramatically in the near future such as malabsorption, pregnancy, malignancy
* For Normal: BMI>30, BP > 140/90 , LDL > 130.
* For Diabetes: BP> 135/85, A1C> 8%. LDL > 100.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient with diabetes or healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2007-04-25 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Carotid intima media measurement change | 2 years
  To describe carotid intima media measurement change over 2 year period in normal individuals compared to individuals with well controlled diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Larsen, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided